CLINICAL TRIAL: NCT07360106
Title: A Proof-of-Concept Study to Assess the Efficacy of Symprove Probiotics in Managing Persistent Gastrointestinal Symptoms in Adult Coeliac Disease Patients in Histological Remission
Brief Title: Efficacy of Symprove Probiotics in Coeliac Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH23479
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Coeliac Disease; Probiotic; Gluten
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open-label, proof-of-concept study evaluating the efficacy of Symprove probiotics in managing persistent gastrointestinal symptoms in adult coeliac disease patients in histological remission. All participants will receive daily Symprove supplementation for 3 months, with assessments at baseline and monthly intervals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Symprove Probiotic (Experimental): All participants will receive a daily oral dose of 70 mL Symprove probiotic supplement for 3 months, with an optional fourth month contingent on completion of all study assessments at month 3. Symprove is a gluten-free, dairy-free probiotic formulation containing live Lactobacillus and Bifidobacterium strains. Participants will self-administer the probiotic daily at home. This is a single-arm, open-label, proof-of-concept study.
  Interventions: Dietary Supplement: Symprove Probiotic

INTERVENTIONS:
Dietary Supplement: Symprove Probiotic — Symprove is a water-based, multi-strain probiotic food supplement containing live bacteria (Lactobacillus and Bifidobacterium strains). Participants will take 70 mL of Symprove orally once daily for 3 months (90 days total), with an optional fourth month available if participants complete all month-3 assessments. The probiotic will be provided free of charge to participants. Symprove is gluten-free and dairy-free, making it suitable for coeliac disease patients. The intervention aims to rebalance gut microbiota dysbiosis and reduce persistent gastrointestinal symptoms in coeliac disease patients in histological remission.

SUMMARY:
Coeliac Disease (CD) is a lifelong autoimmune condition where eating gluten (a protein found in wheat, barley, and rye) causes damage to the small intestine. It affects around 1 in 100 people. Most individuals feel better and their gut heals after switching to a strict gluten-free diet. However, up to 1 in 5 people with coeliac disease continue to experience unpleasant gut symptoms-such as bloating, pain, and diarrhoea-despite following the diet and having a healed intestine. These ongoing symptoms can be very distressing and impact daily life.

This study investigates whether a food supplement called Symprove, a probiotic drink containing live good bacteria, can help relieve these ongoing symptoms. Scientists believe that in some people with coeliac disease, the community of bacteria in the gut (called the microbiota) becomes unbalanced, even after going gluten-free. This imbalance (known as dysbiosis) may lead to inflammation, irritation, and symptoms similar to irritable bowel syndrome (IBS).

The aim of this study is to test whether Symprove can help correct this imbalance and reduce symptoms. Participants will take Symprove daily and their symptoms, quality of life, and gut bacteria (measured from stool samples) will be monitored over time.

The study hopes to answer three key questions: Can Symprove reduce gut symptoms in people with coeliac disease who are in remission? Does it work by restoring a healthy balance of gut bacteria? Are people with more severe imbalance (dysbiosis) more likely to have symptoms?

If successful, this research could offer a safe, non-drug option to improve life for coeliac patients who continue to suffer symptoms despite avoiding gluten. It could also help suggest that gut bacteria play a role in ongoing symptoms and are a target for future treatment.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-65 years with biopsy-confirmed coeliac disease (CD)

Normal duodenal biopsy (Marsh 0 or Marsh I) within the last 12 months, confirming histological remission

Adherence to a strict gluten-free diet (GFD) for at least 6 months

Persistent gastrointestinal (GI) symptoms for at least 6 months despite adherence to GFD and histological remission

Ability to provide written informed consent

Exclusion Criteria:

Active gluten ingestion or non-adherence to a gluten-free diet

Use of antibiotics within the past 3 months

Use of probiotics within the past 3 months

Known comorbidities affecting gastrointestinal function (e.g., Crohn's disease, ulcerative colitis, irritable bowel syndrome with severe diarrhea, or other significant gastrointestinal disorders)

Pregnancy or lactation

Inability to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Gastrointestinal Symptom Scores | Assessed monthly at baseline, Month 1, Month 2, and Month 3
  Clinically significant reduction in gastrointestinal (GI) symptom scores, defined as a reduction of 50 points or more on validated GI symptom assessment scales (such as GSRS-IBS: Gastrointestinal Symptom Rating Scale - Irritable Bowel Syndrome) from baseline. The GSRS-IBS assesses gastrointestinal symptoms including bloating, abdominal pain, diarrhea, and other bowel-related symptoms. A 50-point reduction is considered clinically meaningful. Higher scores indicate worse symptoms, so a reduction indicates improvement.
  Unit of Measure:
  GSRS-IBS total score (continuous variable)

SECONDARY OUTCOMES:
Change in Quality of Life (EQ-5D Scores) | Assessed at baseline and Month 3 (change from baseline to 3 months)
  Quality of life will be measured using the EQ-5D questionnaire, a standardized instrument that assesses five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level scale, and responses are converted into a single index score representing overall health status. The change in EQ-5D index score from baseline (prior to intervention) to 3 months post-intervention will be calculated. Higher scores indicate better health-related quality of life.
  Unit of Measure: EQ-5D index score (continuous variable)
Change in Gut Microbiota Diversity | Assessed at baseline (Month 0) and Month 3
  Changes in gut microbial diversity measured through stool sample analysis using 16S rRNA gene sequencing.
  Gut microbial diversity will be assessed through stool sample analysis using 16S rRNA gene sequencing. Diversity will be quantified using standard ecological metrics. The outcome is the change in gut microbiota diversity from baseline (Month 0) to Month 3. Higher diversity is generally associated with improved gut health.
  Unit of Measure: Diversity indices (e.g. observed species count)

CONTACTS AND LOCATIONS:
Overall Officials: David S Sanders, MBChB, MD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie published results will be made available to researchers upon reasonable request following completion of the trial and publication of the main findings. Data will be stored securely and released only with appropriate approvals, in accordance with the Data Protection Act 2018 and Sheffield Teaching Hospitals NHS Trust policies. Requests for access may come from both internal and external research collaborators, and all IPD will be stripped of direct patient identifiers prior to sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Once main finding and results have been published
Access Criteria: Applications for access will be assessed by the CI and investigator team.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-10-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT07360106/Prot_SAP_000.pdf
  • Informed Consent Form (2025-10-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT07360106/ICF_001.pdf